CLINICAL TRIAL: NCT02154282
Title: iPod Games in Hepatic Encephalopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jasmohan Bajaj, MD, Hunter Holmes Mcguire Veteran Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAJAJ0013
Record Dates: First submitted 2014-05-27; First posted 2014-06-03 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Hepatic Encephalopathy; Cirrhosis
Keywords: hepatic encephalopathy; covert hepatic encephalopathy; cirrhosis
MeSH Terms: conditions — Hepatic Encephalopathy; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ipod games (Experimental): Administered ipod games with cognitive testing before and after
  Interventions: Behavioral: ipod games

INTERVENTIONS:
Behavioral: ipod games — Patients will be given ipod games for 4 weeks and tested in related and unrelated cognitive measures

SUMMARY:
To see if using ipod games can improve mental functioning

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis proven by biopsy, radiology or endoscopy
* Age 18-70
* Able to give informed consent
* Cognitive dysfunction defined by impaired performance on standard cognitive tests

Exclusion Criteria:

* Illicit drug or alcohol use within 3 months
* Trans-jugular intra-hepatic porto-systemic shunt (TIPS) placement
* Need for psychoactive medications apart from continuous anti-depressants or methadone
* Any focal neurological deficit or neuro-muscular disease
* Inability to function with an iPod
* Inability to understand English

For MRI: inability to perform brain MRI is an exclusion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Improvement in cognitive test performance with iPod games | 8 weeks
  improvement in cognitive performance on a battery of cognitive tests (Psychometric Hepatic Encephalopathy Score, Inhibitory Control test and Verbal Learning) after iPod tests

SECONDARY OUTCOMES:
Improvement in health-related quality of life | 8 weeks
  Sickness Impact Profile will be used before and after the treatment
Improvement in brain MRI parameters | 4 weeks
  change in detailed imaging parameters related to diffusion tensor imaging, resting state and voxel-based morphometry

CONTACTS AND LOCATIONS:
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, Virginia, United States